CLINICAL TRIAL: NCT02931942
Title: The Changing Over Time of Ascorbic Acid After Chemotherapy
Brief Title: Changing Over Time of Ascorbic Acid After Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL53414.068.15/METC152025
Record Dates: First submitted 2016-09-15; First posted 2016-10-13 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Leukemia (Both ALL and AML); Cancer of Lung; Myeloma
Keywords: AA
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Lung Neoplasms; Neoplasms, Plasma Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — peripheral blood on AA level and blood count
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- A: Acute leukemia: Patients that will receive intensive clinical chemotherapy for acute leukemia or high risk myelodysplasia (RAEB2) Blood withdrawn 5-7 x
  Interventions: Other: blood withdrawn
- B: Autologous transplantation: Patients that will receive high dose chemotherapy and autologous stem cell rescue for varies hematological malignancies Blood withdrawn 5-7 x
  Interventions: Other: blood withdrawn
- C: controls: Healthy controls, found amongst family members of patients of group A and B Blood withdrawn 5-7 x
  Interventions: Other: blood withdrawn
- D: lung cancer: Patients that will receive relatively mild immunosuppressive chemotherapy for lung cancer, that will mostly be in the outpatient setting Blood withdrawn 5-7 x
  Interventions: Other: blood withdrawn
- E: colon cancer: Patients that will receive relatively mild immunosuppressive chemotherapy for colon cancer, that will mostly be in the outpatient setting and mostly adjuvant Blood withdrawn 5-7 x
  Interventions: Other: blood withdrawn
- F: controls: Healthy controls, found amongst family members of patients of group D and E Blood withdrawn 5-7 x
  Interventions: Other: blood withdrawn

INTERVENTIONS:
Other: blood withdrawn — venous blood sampling

SUMMARY:
Rationale: Recent studies showed that ascorbic acid (AA) stimulates proliferation and maturation of T lymphocytes and NK cells. Chemotherapy results in depletion of those cells and thereby an increased infection rate. A pilot study showed low levels of AA in the plasma of several patients after chemotherapy for hematological malignancies. AA suppletion could be beneficial to the recovery of the immune system in these patients. But before an intervention study can be undertaken, further understanding of changing over time of AA levels and the relationship with the immune status after chemotherapy is necessary.

Objective: The aim of this pilot study is to evaluate the changing over time of AA levels in plasma and in leukocytes before and during chemotherapy treatment for several different groups of patients and compare that to healthy controls. In this way we want to identify the patients were further interventions could be useful and use the data in the development of an intervention study for power calculations and to identify the primary endpoint.

Study design: observational study

Study population: There will be 6 different groups of participants in the study: two groups of patients that receive clinical intensive chemotherapy (acute leukemia and high dose chemotherapy with autologous stem cell rescue), two groups of patients that receive relatively mild chemotherapy in outpatient setting (colon cancer and lung cancer) and two control groups. All participants will be adults and recruited at the MUMC+. In total there will be 150 participants.

Main study parameters/endpoints: Influence of chemotherapy on AA levels in plasma and in leukocytes.

DETAILED DESCRIPTION:
Rationale: Recent studies showed that ascorbic acid (AA) stimulates proliferation and maturation of T lymphocytes and NK cells. Chemotherapy results in depletion of those cells and thereby an increased infection rate. A pilot study showed low levels of AA in the plasma of several patients after chemotherapy for hematological malignancies. AA suppletion could be beneficial to the recovery of the immune system in these patients. But before an intervention study can be undertaken, further understanding of changing over time of AA levels and the relationship with the immune status after chemotherapy is necessary.

Objective: The aim of this pilot study is to evaluate the changing over time of AA levels in plasma and in leukocytes before and during chemotherapy treatment for several different groups of patients and compare that to healthy controls. In this way we want to identify the patients were further interventions could be useful and use the data in the development of an intervention study for power calculations and to identify the primary endpoint.

Study design: observational study

Study population: There will be 6 different groups of participants in the study: two groups of patients that receive clinical intensive chemotherapy (acute leukemia and high dose chemotherapy with autologous stem cell rescue), two groups of patients that receive relatively mild chemotherapy in outpatient setting (colon cancer and lung cancer) and two control groups. All participants will be adults and recruited at the MUMC+. In total there will be 150 participants.

Main study parameters/endpoints: Influence of chemotherapy on AA levels in plasma and in leukocytes.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

If participants really have a lack of AA after chemotherapy, AA supplementation could be beneficial for the immune recovery in many future patients on chemotherapy. However, the participants cannot benefit yet, because this study does not interfere with current clinical practice. The risks associated with participation in this study are low. Venous blood sampling is performed by skilled and experienced laboratory technicians. For the study, only a small amount of blood, 5 to 7 times 17 ml is needed. Therefore no harm can be expected. Blood withdrawal could result in a hematoma, but this is usually not harmful. Bleedings from the blood withdrawal are usually negligible.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* written informed consent
* Require chemotherapy and will start this treatment in less than 1 month after registration for any of the following diseases:

  * Acute leukemia or high risk myelodysplasia (RAEB2)
  * Hematological disease requiring autologous stem cell transplantation after chemotherapy
  * Lung cancer
  * Colon cancer
* Or family member of a participant (without malignancy or chemotherapy)

Exclusion Criteria:

* recent (<1 month ago) chemotherapy
* kidney failure requiring dialysis
* life expectancy < 1 month
* use of immunosuppressive medication other than chemotherapy and corticosteroids
* active vitamin C suppletion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Like explained before, there will be 6 different groups of participants:
  1. Patients that will receive intensive clinical chemotherapy for acute leukemia or high risk myelodysplasia (RAEB2)
  2. Patients that will receive high dose chemotherapy and autologous stem cell rescue for varies hematological malignancies
  3. Patients that will receive relatively mild immunosuppressive chemotherapy for lung cancer, that will mostly be in the outpatient setting
  4. Patients that will receive relatively mild immunosuppressive chemotherapy for colon cancer, that will mostly be in the outpatient setting and mostly adjuvant
  5. Healthy controls, found amongst family members of patients of group 1 and 2
  6. Healthy controls, found amongst family members of patients of group 3 and 4
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
AA level in leukocytes | Baseline to week 4
  change in AA level during chemotherapy

SECONDARY OUTCOMES:
AA level in plasma | Baseline, week 1, week 2, week 3, week 4, week 8
AA level in leukocytes | Baseline to week 1, to week 3, to week 3 and to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Bos, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- MUMC+, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No